CLINICAL TRIAL: NCT03940469
Title: Comparison Between Dexmedetomidine Versus Dexamethasone With Levobupivacaine in Ultrasound Guided Interscalene Block During Shoulder Arthroscopy: A Randomized Controlled Study
Brief Title: Dexmedetomidine Versus Dexamethasone With Levobupivacaine in Interscalene Block
Acronym: IBBB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Mamdoh Elsayed Lotfy (Unknown); Osama Abdallah Elsharkawy (Unknown); Basma Abdelhamid Fathy (Unknown)
Responsible Party: Principal Investigator, ashraf magdy eskandr, Assistant Professor of Anesthesia, ICU, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Interscalene Dexmedetomidine
Record Dates: First submitted 2019-04-10; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Analgesia; Postoperative Complications
Keywords: Dexmedetomidine; Dexamethasone; Interscalene
MeSH Terms: conditions — Postoperative Complications | interventions — Sodium Chloride; Saline Solution; Calcium Dobesilate; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: three groups 20 each, Group C received 35ml levobupivacaine+2ml normal saline under ultrasound guided interscalene block. Group H received 35ml levobupivacaine+8mg dexamethasone under ultrasound guided interscalene block. Group D received 35ml levobupivacaine+100umg dexmedetomidine+1ml normal saline.
Who Masked: Participant, Outcomes Assessor
Masking Description: both the patients and the observer were blind to the treatment groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Placebo Comparator): received 35ml levobupivacaine+2ml normal saline under ultrasound guided interscalene block.
  Interventions: Drug: Saline
- Dexamethasone group (Active Comparator): received 35ml levobupivacaine+8mg dexamethasone
  Interventions: Drug: Dexamethasone Injection
- Dexmeteomidine group (Active Comparator): received 35ml levobupivacaine+100umg dexmedetomidine+1ml normal saline.
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Saline — 2 ml normal saline
  Other Names: normal saline
  Arms: Control group
Drug: Dexamethasone Injection — 8 mg dexamethasone
  Other Names: dexamethsone
  Arms: Dexamethasone group
Drug: Dexmedetomidine Hydrochloride — 100 microgram dexmedetomidine
  Other Names: dexmedetomidine
  Arms: Dexmeteomidine group

SUMMARY:
The investigators compared between dexamethasone and dexmedetomidine when added to levobupivacaine in the quality and duration of ultrasound-guided interscalene block during shoulder arthroscopy.

DETAILED DESCRIPTION:
Sixty patients were enrolled and divided into three groups 20 each, Group C received 35ml levobupivacaine+2ml normal saline under ultrasound guided interscalene block. Group H received 35ml levobupivacaine+8mg dexamethasone under ultrasound guided interscalene block. Group D received 35ml levobupivacaine+100umg dexmedetomidine+1ml normal saline. The primary outcome was the postoperative pain which was assessed by Visual analog score(VAS), the secondary outcomes were the onset and duration of sensory and motor block, the total amount of analgesic requirement, and blood cortisol level.

ELIGIBILITY:
Inclusion Criteria:

* Sixty healthy patients ASA I-II
* Aged 18-60 years
* Of both sexes
* Scheduled for shoulder arthroscopy using ultrasound interscalene block were enrolled.

Exclusion Criteria:

* Patients with a history of any allergic reactions to levobupivacaine, dexamethasone or α2 agonists
* All patients with hypertension, cardiac, hepatic, renal or pulmonary diseases, - Patients who were under treatment by α2 agonist or antagonists
* Pregnant women
* Psychiatric patients
* Patients with a previous history or clinical evidence of central or peripheral neurological disease
* Coagulopathy or anticoagulant/antiaggregant therapy
* Contralateral phrenic nerve paresis
* Patients who have an infection at the site of the block.
* Every patient who had an anatomical or vascular abnormality in the upper extremity were excluded from this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-03 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in postoperative analgesia | During first 2 days after surgery
  Assessed by measuring severity of pain by visual analog score(score 0 to 10 cm with 0= no pain and 10=worst pain imaginable).

SECONDARY OUTCOMES:
Postoperative analgesic requirement | During first 2 days after surgery
  Total amount of paracetamol required in mg
Hemodynamic parameter | During first 2 days after surgery
  Heart rate
Hemodynamic parameter | During first 2 days after surgery
  Mean arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: mamdouh e lotfy, m.d., Study Director — emeritus professor
Locations (1):
- Ashraf Eskandr, Shibīn al Kawm, Monufia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No